CLINICAL TRIAL: NCT02216916
Title: Phase II Trial of HM781-36B in Patients With Metastatic/Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC) After Failure of or Unfit for Platinum-containing Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0794
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — HM781-36B; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HM781-36B (Experimental)
  Interventions: Drug: HM781-36B

INTERVENTIONS:
Drug: HM781-36B
  Other Names: 45 mg p.o. daily and continuously (28-day treatment as one treatment cycle)

SUMMARY:
Head and neck cancer is the sixth most common cancer and more than 650,000 new cases are diagnosed each year worldwide. About 60% of the HNSCC patients present with unresectable locally advanced disease at diagnosis and treated with multimodality approach. Despite such approach, majority (70%) of patients develop local or/and regional recurrences. Additional 10% of patients present with distant metastasis at diagnosis. Most patients with recurrent or metastatic disease are treated with single agent chemotherapy, combination chemotherapy or targeted therapies.

Despite its public health magnitude, HNSCC in Asian countries has received a limited attention for the drug development and cancer-related research. In fact, HNSCC ranked 7th among men and 10th among women by incidence in China, the largest producer and consumer of tobacco and alcohol. Recently, Chen et al. documented a 1:1:2 subset distribution for cancers of oral cavity, pharynx, and larynx in China, similar to the distribution reported in Korea but quite different from the general distribution of 5:2:3 in whites. Ethnic disparities in HNSCC also include its prognosis and this is partly explained by HPV-active disease ratio and genetic factors. Therefore, there is a strong need for an additional research in patients with HNSCC in Asia.

Epidermal growth factor receptor (EGFR) is often over-expressed, and have been related to poor prognosis in patients with HNSCC. The association between EGFR-activated signaling pathways and tumor cell survival are well documented in many studies. EGFR targeting strategies showed clinical anti-tumor efficacy in patients with HNSCC, especially with monoclonal antibody, cetuximab. In the Extreme study, it was shown that the addition of cetuximab to platinum-5-FU significantly prolonged the median overall survival from 7.4 months to 10.1 months compared to platinum-5FU alone in the first-line setting.

HM781-36B is a irreversible pan-HER inhibitor. In preclinical studies, HM781-36B has much lower IC50 values than gefitinib in cell lines engineered to express EGFRvIII mutations and produces tumor growth inhibition in gefitinib-resistant xenografts. A phase I trial of HM781-36B in patients with advanced solid tumors showed clinically significant anti-tumor activity and a phase II trials of HM781-36B in patients with non-small cell lung cancer and advanced gastric cancer are currently ongoing.

We suggest a phase II trial of HM781-36B in patients with recurrent or metastatic HNSCC who are resistant or ineligible/intolerant to platinum-based chemotherapy. The aim of current trial is to evaluate the antitumor efficacy and safety profile of HM781-36B and to identify biomarker to predict the tumor response to HM781-36B.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of head and neck
2. Age ≥ 20 years
3. ECOG PS 0-1

   * Documented progressive disease after platinum-based (either cisplatin or carboplatin) concurrent chemoradiation including induction chemotherapy for curative aim or
   * Documented progressive disease after platinum-based (either cisplatin or carboplatin) chemotherapy for palliative aim or
   * Ineligible to platinum-based (either cisplatin or carboplatin) chemotherapy or chemoradiation due to decline in renal function and patient's intolerance
4. At least one bidimensionally measurable disease as defined by RECIST ver 1.1
5. Adequate organ function for treatment

   * Absolute neutrophil count (ANC) ≥ 1000cells/mm3
   * Platelets ≥ 100000 cells/mm3
   * Estimated creatinine clearance ≥ 50mL/min, or serum creatinine < 1.5 x institution upper limit of normal
   * Bilirubin ≤ 1.5 x upper limit of normal(ULN)
   * AST(SGOT) ≤ 2.5 x ULN (5.0xULN if hepatic metastases)
   * ALT(SGPT) ≤ 2.5 x ULN (5.0xULN if hepatic metastases)
6. The patient has provided signed informed consent and is amenable to compliance with protocol schedules and testing

Exclusion Criteria:

1. Nasopharyngeal carcinoma
2. Patients who are subjected to local treatment (surgery or radiation)
3. Previous treatment with small molecule EGFR tyrosine kinase inhibitors (Cetuximab is permitted)
4. Three or more previous systemic cytotoxic chemotherapy
5. Any major operation or irradiation within 4 weeks of baseline disease assessment
6. Patients who have received prior systemic chemotherapy, immunotherapy or study drug within 4 weeks
7. Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
8. Patients with uncontrolled CNS metastatic involvement. However, patients with metastatic CNS tumors may participate in this study if the patient is clinically stable not receiving steroid therapy more than 1 week from prior therapy completion (including radiation and/or surgery) to stating the study drug.
9. Patients with known interstitial lung disease (ILD) or presented ILD on screening chest X-ray
10. Congenital long QT syndrome or screening corrected QT interval (QTc) > 470msec
11. Patients with uncontrolled or significant cardiovascular disease (AMI within 12 months, Unstable angina within 6 months, NYHA Class III, IV Congestive heart failure or left ventricular ejection fraction below local institutional lower limit of normal or below 45%, Congenital long QT syndrome, Any significant ventricular arrhythmia, Any uncontrolled second or third degree heart block, Uncontrolled hypertension)
12. Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to study entry.
13. Pregnant or breast-feeding women
14. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2014-08; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Response rate | 28th day of 1st chemotherapy cycle
  Objective Tumor Response will be performed according to the Response Evaluation in Solid Tumor Criteria 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Best Overall Response | 1years
Duration of response | 1years
Progression-Free Survival | 1years
Overall Survival | 1years
Toxicity profile | 1years
  Overall safety profile and toleration of HM781-36B will be characterized by type, frequency, severity (as graded by the NCI CTCAE v4.02), timing and relationship of study therapy of adverse events and laboratory abnormalities. Quantitative variables will be summarized in descriptive terms.
Quality of Life (QoL) | 1years
  Questionnaire
Identification of predictive markers of treatment | 1years
  * To explore KRAS and HER family mutation status in tissue at the end of treatment;
  * To explore the pre- and post-treatment levels of shed proteins/receptors related to HER signaling (possibly to include EGFR and HER-2 receptor extracellular domain (ECD) and E-cadherin);

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Heo SG, Ahn BC, Hong MH, Cho BC, Lim SM, Kim HR. A phase II study of poziotinib in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Cancer Med. 2021 Oct;10(20):7012-7020. doi: 10.1002/cam4.4231. Epub 2021 Sep 16. PMID 34528763